CLINICAL TRIAL: NCT02401308
Title: Randomized Controlled Clinical Trial Comparing Functional Outcomes of Awake vs. Asleep Deep Brain Stimulation (DBS) for Parkinson's Disease
Brief Title: Trial Comparing Functional Outcomes of Awake vs. Asleep Deep Brain Stimulation (DBS) for Parkinson's Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of subject enrollment.
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB # 14BN147
Record Dates: First submitted 2015-03-24; First posted 2015-03-27 (Estimated); Results first posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-09

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Awake DBS Surgery (Active Comparator): Deep brain stimulation surgery: Parkinson's patients undergoing traditional "awake" DBS surgery utilizing microelectrode recordings and intra-operative stimulation
  Interventions: Procedure: Deep Brain Stimulation surgery
- Asleep DBS Surgery (Active Comparator): Deep brain stimulation surgery:Parkinson's patients undergoing DBS surgery under general anesthesia utilizing intraoperative imaging to verify the stereotactic accuracy of DBS electrodes placement at the time of surgery.
  Interventions: Procedure: Deep Brain Stimulation surgery

INTERVENTIONS:
Procedure: Deep Brain Stimulation surgery — Deep Brain Stimulation surgery: awake vs. asleep
  Other Names: DBS

SUMMARY:
The purpose of the proposed study is to demonstrate that the functional outcomes of DBS surgery utilizing the "asleep" technique are not inferior to those reported for traditional "awake" DBS technique.

DETAILED DESCRIPTION:
Traditional DBS is performed without general anesthesia with the patient awake. Local anesthetic is used to numb the skin and tissue where the incision is made, and the patients are given mild sedatives to alleviate anxiety and discomfort. Parkinson's patients need to be off their medications during awake DBS in order to obtain single-unit cellular recordings to locate and map the desired target. The process of electrophysiological mapping can result in multiple brain penetrations during lead placement, and the entire procedure may last anywhere from 4-6 hours on average. The concept of being awake during brain surgery and being off medications are significant concerns for some patients. In addition, it is widely recognized that microelectrode recording increases the risk of hemorrhage during DBS surgery.

Recently, there has been increasing interest in performing DBS under general anesthesia, where the stimulated targets are located anatomically (i.e. on MRI) rather than physiologically via microelectrode recordings. This technology has been termed "asleep" DBS and is performed with the patient under general anesthesia. Intraoperative imaging is utilized to verify the stereotactic accuracy of DBS electrodes placement at the time of surgery. Because stereotactic accuracy (and surgical safety) is the surgical endpoint, there is no need for the patient to be off medication and awake during the procedure.

Traditional DBS is performed without general anesthesia with the patient awake. Local anesthetic is used to numb the skin and tissue where the incision is made, and the patients are given mild sedatives to alleviate anxiety and discomfort. Parkinson's patients need to be off their medications during awake DBS in order to obtain single-unit cellular recordings to locate and map the desired target. The process of electrophysiological mapping can result in multiple brain penetrations during lead placement, and the entire procedure may last anywhere from 4-6 hours on average. The concept of being awake during brain surgery and being off medications are significant concerns for some patients. In addition, it is widely recognized that microelectrode recording increases the risk of hemorrhage during DBS surgery.

The safety and efficacy of the two approaches to DBS surgery have been equivalent, and we are at a position of equipoise with regard to what to offer to patients. To date, there have been no randomized, controlled clinical trials comparing the efficacy and functional outcomes of the two DBS methods. After informed consent is obtained, the patients will undergo routine DBS pre-operative evaluation and diagnostic testing. This includes a pre-operative 3T-MRI with and without gadolinium as well as pre-operative medical clearance by the patient's PCP or general practitioner and/or other medical specialist if necessary. They will also receive a baseline clinical evaluation including both motor function (Unified Parkinson's Disease Rating Scale on and off antiparkinsonian medication) and quality of life (Parkinson's disease Questionnaire-39) if not already completed as part of the routine DBS candidacy evaluation within 2 months of surgery. Patients who elect to participate in this trial will undergo a routine pre-operative neurocognitive evaluation consisting of the following routine evaluative tests: Wechsler Test of Adult Reading, Mattis Dementia Rating Scale 2nd Edition, Wechsler Abbreviate Scale of Intelligence 2nd Edition; Wechsler Memory Scale 3rd edition, Digit Span, Stroop Neuropsychological Screening Test, Trail Making Test, Wisconsin Card Sorting Test, Controlled Oral Word Association Test, Animal Naming, Boston Naming Test, Wechsler Memory Scale 4th Edition, Logical Memory, Hopkins Verbal Learning Test - Revised, Brief Visuospatial Memory Test - Revised, Hooper visual Organization Test, Judgment of Line Orientation, Beck Depression Inventory, Beck Anxiety Inventory, Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease, Apathy Evaluation Scale; Epworth Sleepiness Scale, The subjects will then be randomized to 2 groups by using random numbers in an envelope system. We anticipate that 120 total patients will need to be enrolled in this pilot study (60 awake, 60 asleep), and thus the numbers 1-120 will be placed in envelopes. An odd number will correspond to the awake DBS procedure, and an even number will indicate an asleep DBS procedure.

The purpose of the proposed study is to demonstrate that the functional outcomes of the "asleep" technique are not inferior to those reported for traditional "awake" DBS technique. The primary data points for this study will include six month functional outcomes using accepted metrics for Parkinson's disease, including both motor function (Unified Parkinson's Disease Rating Scale [UPDRS] obtained in the medication "on" and medication "off" states) and quality of life (Parkinson's Disease Questionnaire-39). The null hypothesis is that asleep DBS results in inferior UPDRS-III scores at 6-months after surgery. Our secondary aim will be to evaluate any cognitive changes associated with DBS surgery selection (awake vs. asleep) in PD patients. Current standard of care for patient selection in DBS focuses primarily on the evaluation of motor symptoms and currently there is no guidance for how a patients' DBS surgery selection (awake vs. asleep) would impact on subsequent neurocognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease per Queens Square criteria
* Appropriate DBS candidate for multi-disciplinary team consensus
* Age 18 - 85 years of age
* Motor skills allowing for capability to complete evaluations
* Medically cleared for undergoing anesthesia and DBS surgery

Exclusion Criteria:

* Dementia per DSM-V criteria
* Medical or other condition precluding MRI
* History of supraspinal CNS disease other than PD
* Alcohol use of more than 4 drinks per day
* Pregnancy
* History of suicide attempt
* Currently uncontrolled clinically significant depression (BDI>20)
* History of schizophrenia, delusions, or currently uncontrolled visual hallucinations

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-01-15 (Actual); Primary Completion 2015-10-05 (Actual); Study Completion 2015-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco A Ponce, MD, Principal Investigator — Barrow Neurological Institute / St. Joseph's Hosptial and Medical Center
Locations (1):
- Barrow Neurological Institute / St. Joseph's Hospital & Medical Center, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ostrem JL, Galifianakis NB, Markun LC, Grace JK, Martin AJ, Starr PA, Larson PS. Clinical outcomes of PD patients having bilateral STN DBS using high-field interventional MR-imaging for lead placement. Clin Neurol Neurosurg. 2013 Jun;115(6):708-12. doi: 10.1016/j.clineuro.2012.08.019. Epub 2012 Sep 1. PMID 22944465
- [Background] Nakajima T, Zrinzo L, Foltynie T, Olmos IA, Taylor C, Hariz MI, Limousin P. MRI-guided subthalamic nucleus deep brain stimulation without microelectrode recording: can we dispense with surgery under local anaesthesia? Stereotact Funct Neurosurg. 2011;89(5):318-25. doi: 10.1159/000330379. Epub 2011 Sep 15. PMID 21921673
- [Background] Harries AM, Kausar J, Roberts SA, Mocroft AP, Hodson JA, Pall HS, Mitchell RD. Deep brain stimulation of the subthalamic nucleus for advanced Parkinson disease using general anesthesia: long-term results. J Neurosurg. 2012 Jan;116(1):107-13. doi: 10.3171/2011.7.JNS11319. Epub 2011 Oct 14. PMID 21999316
- [Background] Weaver FM, Follett K, Stern M, Hur K, Harris C, Marks WJ Jr, Rothlind J, Sagher O, Reda D, Moy CS, Pahwa R, Burchiel K, Hogarth P, Lai EC, Duda JE, Holloway K, Samii A, Horn S, Bronstein J, Stoner G, Heemskerk J, Huang GD; CSP 468 Study Group. Bilateral deep brain stimulation vs best medical therapy for patients with advanced Parkinson disease: a randomized controlled trial. JAMA. 2009 Jan 7;301(1):63-73. doi: 10.1001/jama.2008.929. PMID 19126811
- [Background] Pezeshkian P, DeSalles AA, Gorgulho A, Behnke E, McArthur D, Bari A. Accuracy of frame-based stereotactic magnetic resonance imaging vs frame-based stereotactic head computed tomography fused with recent magnetic resonance imaging for postimplantation deep brain stimulator lead localization. Neurosurgery. 2011 Dec;69(6):1299-306. doi: 10.1227/NEU.0b013e31822b7069. PMID 21725253
- [Background] Papanastassiou V, Rowe J, Scott R, Silburn P, Davies L, Aziz T. Use of the Radionics Image Fusiontrade mark and Stereoplantrade mark programs for target localization in functional neurosurgery. J Clin Neurosci. 1998 Jan;5(1):28-32. doi: 10.1016/s0967-5868(98)90197-7. PMID 18644283
- [Background] Alexander E 3rd, Kooy HM, van Herk M, Schwartz M, Barnes PD, Tarbell N, Mulkern RV, Holupka EJ, Loeffler JS. Magnetic resonance image-directed stereotactic neurosurgery: use of image fusion with computerized tomography to enhance spatial accuracy. J Neurosurg. 1995 Aug;83(2):271-6. doi: 10.3171/jns.1995.83.2.0271. PMID 7616273
- [Background] Kooy HM, van Herk M, Barnes PD, Alexander E 3rd, Dunbar SF, Tarbell NJ, Mulkern RV, Holupka EJ, Loeffler JS. Image fusion for stereotactic radiotherapy and radiosurgery treatment planning. Int J Radiat Oncol Biol Phys. 1994 Mar 30;28(5):1229-34. doi: 10.1016/0360-3016(94)90499-5. PMID 8175410

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Awake DBS Surgery | Asleep DBS Surgery
Started | 0 | 1
Completed | 0 | 0
Not Completed | 0 | 1
Not completed — Study was terminated by the PI due to lack of enrollment. | 0 | 1

BASELINE CHARACTERISTICS:
Population: Study was terminated due to lack of enrollment. Only 1 subject was enrolled. No analysis was completed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Awake DBS Surgery | Asleep DBS Surgery | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Functional Outcomes
Description: Motor function outcomes using accepted metrics for Parkinson's disease - the Unified Parkinson's Disease Rating Scale [UPDRS] obtained in 3 states:
  1. medication "off" / device "on".
  2. Medication "off" / device "off"
  3. medication "on" / device "on"
Time Frame: 6 months post-operatively
Population: Study was terminated due to lack of enrollment. No analysis was completed.
Arm/Group | Awake DBS Surgery | Asleep DBS Surgery
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Neurocognitive Function
Description: Neurocognitive evaluation consisting of the following routine evaluative tests: Wechsler Test of Adult Reading, Mattis Dementia Rating Scale 2nd Edition, Wechsler Abbreviate Scale of Intelligence 2nd Edition; Wechsler Memory Scale 3rd edition, Digit Span, Stroop Neuropsychological Screening Test, Trail Making Test, Wisconsin Card Sorting Test, Controlled Oral Word Association Test, Animal Naming, Boston Naming Test, Wechsler Memory Scale 4th Edition, Logical Memory, Hopkins Verbal Learning Test - Revised, Brief Visuospatial Memory Test - Revised, Hooper visual Organization Test, Judgment of Line Orientation, Beck Depression Inventory, Beck Anxiety Inventory, Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease, Apathy Evaluation Scale; Epworth Sleepiness Scale.
Time Frame: 6 months post-operatively
Population: Study was terminated due to lack of enrollment. No analysis was completed.
Arm/Group | Awake DBS Surgery | Asleep DBS Surgery
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Quality of Life
Description: Parkinson's Disease Questionnaire-39 to evaluate the patient's assessment of their quality of life following DBS surgery
Time Frame: 6 months post-operatively
Population: Study was terminated due to lack of enrollment. No analysis was completed.
Arm/Group | Awake DBS Surgery | Asleep DBS Surgery
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Per protocol, participants were to be followed for 6 months post surgery.
Description: Only 1 subject was enrolled and he was randomized to the asleep arm. Therefore, there were no subjects at risks for AEs in the Awake Arm.
Arm/Group | Awake DBS Surgery | Asleep DBS Surgery
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1

LIMITATIONS AND CAVEATS:
This trial was terminated without meeting the objectives. One out of the planned 120 participants was enrolled. There was no analysis completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes